CLINICAL TRIAL: NCT06399718
Title: BOTOX® (onabotulinumtoxinA) for the Reduction of Masseter Muscle Prominence: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study
Brief Title: A Study to Assess BOTOX Injections for the Change of Masseter Muscle Prominence in Adult Participants
Acronym: MMP US P3 417
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: M21-417
Record Dates: First submitted 2024-05-01; First posted 2024-05-06 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Masseter Muscle Prominence
Keywords: BOTOX; OnabotulinumtoxinA; Masseter Muscle Prominence
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Double-Blind Period: BOTOX (Experimental): Participants will receive BOTOX injections across both the right and left masseter muscle on Day 1.
  Interventions: Drug: BOTOX
- Double-Blind Period: Placebo (Placebo Comparator): Participants will receive placebo injections across both the right and left masseter muscle on Day 1.
  Interventions: Drug: Placebo
- Open-Label Period: BOTOX (Experimental): Participants who are eligible for re-treatment will receive BOTOX injections on either the Day 180, 210, 240, or 270 visit and will be followed for up to 6 months.
  Interventions: Drug: BOTOX

INTERVENTIONS:
Drug: BOTOX — Intramuscular Injections
  Other Names: OnabotulinumtoxinA
  Arms: Double-Blind Period: BOTOX; Open-Label Period: BOTOX
Drug: Placebo — Intramuscular Injections
  Arms: Double-Blind Period: Placebo

SUMMARY:
The masseter muscle is one of the muscles in the lower face used for chewing. The prominence of the masseter muscle can appear as a widened lower face which some individuals deem as aesthetically undesirable and can be treated by selectively weakening the masseter muscles with small quantities of botulinum toxin. The purpose of this study is to assess how safe and effective injection of onabotulinumtoxinA (BOTOX) is in adult participants with Masseter Muscle Prominence (MMP).

BOTOX is being investigated for the treatment of Muscle Masseter Prominence. In Period 1, participants are placed in 1 of 2 groups, called treatment arms. Each group receives a different treatment, placebo or BOTOX. There is a 1 in 4 chance that participants will be assigned to placebo. In Period 2, eligible participants can receive an optional open-label retreatment of BOTOX. Approximately 200 adult participants with MMP will be enrolled in the study at approximately 20 sites in the United States.

Participants will receive intramuscular injections across both the right and left masseter muscle of either BOTOX or placebo on Day 1. Participants who are eligible for re-treatment will be given a BOTOX injection on either the Day 180, 210, 240, or 270 visit and will be followed up for up to 6 months.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular monthly visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, checking for side effects, and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Participant meets the following criteria:

  * Bilateral Grade 4 or Grade 5 Masseter Muscle Prominence (MMP) (identical grades for left and right sides of the face), as determined by the investigator using the Masseter Muscle Prominence Scale (MMPS).
  * Bilateral Grade 4 or Grade 5 MMP (identical grades for left and right sides of the face), as determined by the participant using the Masseter Muscle Prominence Scale - Participant (MMPS-P).
  * Investigator and participant scoring of MMPS and MMPS-P must be the same.
* Body mass index (BMI) ≤ 30 kg/m^2 using the calculation: BMI = weight (kg)/height (m)^2.

Exclusion Criteria:

* Excess lower facial fat, jowling, loose or lax skin in lower face, or parotid gland prominence that could interfere with MMPS or MMPS-P grading.
* Asymmetry of left and right sides of the face that could prevent identical MMPS or MMPS-P grading on both sides of the face.
* History of or current temporomandibular disorder (TMJD), or presence of signs/symptoms of possible TMJD.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2024-04-30 (Actual); Primary Completion 2025-11-10 (Actual); Study Completion 2025-11-10 (Actual)

PRIMARY OUTCOMES:
Composite Achievement of MMP Severity Improvement and at Least a 2-Grade Improvement from Baseline by Both Investigator-Rated MMPS and Participant-Rated MMPS-P | Day 90
  The investigator and participant each assessed the participant's Masseter Muscle Prominence (MMP) using the Masseter Muscle Prominence Scale (MMPS) and the Masseter Muscle Prominence Scale-Participant (MMPS-P), respectively. Both are a 5-point masseter muscle severity scale with grades ranging from 1 (minimal/not at all noticeable) to 5 (very marked/extremely noticeable).
Number of Participants with Adverse Events (AEs) | Baseline to Day 360
  An AE is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.

SECONDARY OUTCOMES:
Percentage of Participants who Responded as "Very satisfied" or "Satisfied" on the Lower Facial Shape Questionnaire - Treatment Satisfaction Assessment (LFSQ-TXSAT) | Day 90
  The LFSQ-TXSAT measures satisfaction with the effect of treatment using a 5-point scale ranging from 'Very satisfied' to 'Very dissatisfied.'
Percentage of Participants who Responded as "Not at all bothered" or "A little bothered" on the Bother Impact Assessment for Masseter Muscle Prominence (BIA-MMP) | Day 90
  The BIA-MMP is a single item evaluation of how bothered the participant is by the appearance of their lower face using a 5-point scale from 'Not at all bothered' to 'Extremely bothered.'
Change from Baseline in Lower Facial Shape Questionnaire-Impact Assessment (LFSQ-IA) Summary Score | Baseline to Day 90
  The LFSQ-IA measures psychosocial impact due to the appearance of the lower face. The LFSQ-IA summary score ranges from '0 (best)' to '24 (worst).'
Percentage of Participants Achieving Investigator-Rated MMPS Improvement Over Time | Baseline to Day 360
  The investigator assessed the participant's MMP using the MMPS, a 5-point masseter muscle severity scale with grades ranging from 1 (minimal) to 5 (very marked).
Percentage of Participants Achieving Participant-Rated MMPS-P Improvement Over Time | Baseline to Day 360
  The investigator assessed the participant's MMP using the MMPS-P, a 5-point masseter muscle severity scale with grades ranging from 1 (not at all noticeable) to 5 (extremely noticeable).

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (20):
- United States (20):
  - Westside Aesthetics /ID# 248232, Los Angeles, California
  - Private Practice - Dr. Steven G. Yoelin /ID# 268046, Newport Beach, California
  - Pacific Clinical Innovations /ID# 248231, Vista, California
  - Sherber + RAD /ID# 248894, Washington D.C., District of Columbia
  - Steven Fagien MD Aesthetic Eyelid Plastic Surgery /ID# 248478, Boca Raton, Florida
  - Skin Research Institute LLC /ID# 248230, Coral Gables, Florida
  - Kavali Plastic Surgery and Skin Renewal Center /ID# 248480, Atlanta, Georgia
  - DeNova Research /ID# 248237, Chicago, Illinois
  - DelRicht Research /ID# 250313, Baton Rouge, Louisiana
  - Etre Cosmetic Dermatology and Laser Center /ID# 248229, New Orleans, Louisiana
  - Aesthetic Center at Woodholme /ID# 248481, Baltimore, Maryland
  - Michigan Center for Research Corporation /ID# 249145, Clinton Township, Michigan
  - Skin Specialists /ID# 248233, Omaha, Nebraska
  - Laser & Skin Surgery Center of New York /ID# 248479, New York, New York
  - Luxurgery /ID# 248236, New York, New York
  - The Practice of Brian S. Biesman MD PLLC /ID# 248226, Nashville, Tennessee
  - Sherman Aesthetic Center /ID# 248482, Nashville, Tennessee
  - Westlake Dermatology & Cosmetic Surgery - Westlake /ID# 249875, Austin, Texas
  - DermResearch Inc. /ID# 248227, Austin, Texas
  - Austin Institute for Clinical Research at SBA Dermatology /ID# 248228, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M21-417